CLINICAL TRIAL: NCT00227695
Title: Comparing Two Schedules of Rituximab Maintenance in Rituximab-Responding Patients With Untreated, Chemotherapy Resistant or Relapsed Follicular Lymphoma: A Randomized Phase III Trial
Brief Title: Rituximab in Treating Patients With Follicular Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Swiss Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SAKK 35/03; SWS-SAKK-35/03; EU-20520; CDR0000443594
Record Dates: First submitted 2005-09-26; First posted 2005-09-28 (Estimated); Last update posted 2019-05-15 (Actual); Status verified 2019-05

CONDITIONS: Lymphoma
Keywords: stage I grade 1 follicular lymphoma; stage I grade 2 follicular lymphoma; stage I grade 3 follicular lymphoma; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; contiguous stage II grade 1 follicular lymphoma; contiguous stage II grade 2 follicular lymphoma; contiguous stage II grade 3 follicular lymphoma; noncontiguous stage II grade 1 follicular lymphoma; noncontiguous stage II grade 2 follicular lymphoma; noncontiguous stage II grade 3 follicular lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Follicular | interventions — Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A: Rituximab every 2 months x4 (Active Comparator): Rituximab 375 mg/m2 every 2 months x4
  Interventions: Biological: rituximab
- Arm B: Rituximab (5 years) (Active Comparator): Rituximab 375 mg/m2 every 2 months for 5 years or until PD, relapse or unacceptable toxicity
  Interventions: Biological: rituximab

INTERVENTIONS:
Biological: rituximab — comparing two maintenance schedules of Rituximab
  Other Names: MABTHERA

SUMMARY:
RATIONALE: Monoclonal antibodies, such as rituximab, can block cancer growth in different ways. Some block the ability of cancer cells to grow and spread. Others find cancer cells and help kill them or carry cancer-killing substances to them. It is not yet known whether giving rituximab over a short period of time is more effective than giving it over a long period of time in treating follicular non-Hodgkin's lymphoma.

PURPOSE: This randomized phase III trial is studying rituximab to see how well it works when given over a short period of time compared to when given over a long period of time in treating patients with follicular non-Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the efficacy of induction therapy with rituximab followed by short- vs long-term maintenance therapy with rituximab, in terms of event-free survival, in patients with follicular non-Hodgkin's lymphoma.

Secondary

* Compare the safety of these regimens in these patients.
* Compare the pharmaeconomical aspects of these regimens in these patients.
* Compare the evolution of immunologic competence in patients treated with these regimens.

OUTLINE: This is a randomized, multicenter study.

* Induction therapy: Patients receive rituximab IV weekly in weeks 1-4 and undergo restaging between weeks 11-13. Patients with stable disease or progressive disease are taken off study. Patients achieving partial or complete response are stratified according to prior treatment status (untreated* vs treated with or without anti-CD20 therapy), presence of bulky disease** at study entry (yes vs no), and participating center. Patients are then randomized to 1 of 2 maintenance treatment arms.

NOTE: *Patients treated with radiotherapy only are considered as therapy-naïve.

NOTE: **Defined as a mass or lymph node conglomerate ≥ 5 cm diameter.

* Maintenance therapy: Patients start maintenance therapy within 7 days of randomization.

  * Arm I: Patients receive rituximab IV every 2 months for 4 treatments.
  * Arm II: Patients receive rituximab IV every 2 months for up to 5 years in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed every 3 months until disease progression or relapse and then annually for up to 10 years after randomization.

PROJECTED ACCRUAL: A total of 270 patients will be accrued for this study within 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed follicular lymphoma

  * Grade 1, 2, 3a, or 3b disease by WHO staging system
* CD20-positive by immunohistochemistry
* Previously untreated disease OR meets 1 of the following criteria for response to prior treatment:

  * Chemotherapy-resistant disease
  * Relapsed or progressive disease
  * Stable disease

    * At least 12 weeks since prior systemic treatment
* At least 1 bidimensionally measurable lesion ≥ 11 mm by CT scan or MRI
* No transformation to high-grade lymphoma secondary to low-grade follicular lymphoma
* No prior or current CNS disease (i.e., CNS lymphoma or lymphomatous meningosis) NOTE: A new classification scheme for adult non-Hodgkin's lymphoma has been adopted by PDQ. The terminology of "indolent" or "aggressive" lymphoma will replace the former terminology of "low", "intermediate", or "high" grade lymphoma. However, this protocol uses the former terminology.

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* WHO 0-2

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* Not specified

Renal

* Not specified

Cardiovascular

* Ejection fraction ≥ 50% by echocardiography or MUGA

Immunologic

* No acute or ongoing infection
* No HIV infection
* No active autoimmune disease

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 12 months after completion of the study treatment
* No uncontrolled diabetes mellitus
* No other medical condition that would preclude study participation
* No other malignancy except nonmelanoma skin cancer or adequately treated carcinoma in situ of the cervix
* No other condition (e.g., geographic proximity) that would preclude study compliance and follow-up

PRIOR CONCURRENT THERAPY:

Biologic therapy

* See Radiotherapy
* Prior rituximab allowed

Chemotherapy

* See Disease Characteristics

Endocrine therapy

* More than 4 weeks since prior regular administration of corticosteroids

  * Dose equivalent to ≤ 20 mg/day prednisone allowed for conditions other than lymphoma or lymphoma-related symptoms
* No concurrent corticosteroids for prevention or treatment of side effects except acute life-threatening side effects

Radiotherapy

* Prior radiolabeled anti-CD20 therapy (administered alone or in combination with cytostatic drugs) allowed provided patient has achieved partial or complete response after the therapy

  * At least 12 months since prior anti-CD20 therapy

Surgery

* Not specified

Other

* More than 30 days since prior systemic tumor therapy
* More than 30 days since prior participation in another clinical trial
* No other concurrent anticancer therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Actual)
Dates: Start 2004-06-08 (Actual); Primary Completion 2013-05-03 (Actual); Study Completion 2017-12-19 (Actual)

PRIMARY OUTCOMES:
Event-free survival | at 10 years

SECONDARY OUTCOMES:
Progression-free survival | at 10 years
Overall survival | at 10 years
Adverse reactions during and after maintenance treatment | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Christian Taverna, MD, Study Chair — Kantonsspital Münsterlingen; Michele Ghielmini, Prof., Study Chair — IOSI - Ospedale San Giovanni, Bellinzona
Locations (26):
- Clinical Center - Institute of Hematology, São Paulo, Brazil
- Istituto Europeo di Oncologia IEO, Milan, Italy
- Clinical Center Skopje, Skopje, North Macedonia
- Clinical Center of Serbia, Belgrade, Serbia
- NOU - National Institute for Oncology, Bratislava, Slovakia
- South Africa (2):
  - Panorama Medical Centre, Cape Town
  - Sandton Oncology Centre, Johannesburg
- Switzerland (19):
  - Kantonspital Aarau, Aarau
  - Kantonsspital Baden, Baden
  - St. Claraspital AG, Basel
  - Universitaetsspital Basel, Basel
  - Istituto Oncologico della Svizzera Italiana - Ospedale Regionale Bellinzona e Valli, Bellinzona
  - Inselspital Bern, Bern
  - Breitenbach Praxis Dr. Haberthür, Breitenbach
  - Kantonsspital Bruderholz, Bruderholz
  - Kantonsspital Graubuenden, Chur
  - Hopital Cantonal Universitaire de Geneve, Geneva
  - Centre Hospitalier Universitaire Vaudois, Lausanne
  - Kantonsspital, Liestal
  - Istituto Oncologico della Svizzera Italiana, Lugano
  - Hôpital Pourtalès, Neuchâtel
  - Kantonsspital - St. Gallen, Sankt Gallen
  - SpitalSTS AG Simmental-Thun-Saanenland, Thun
  - City Hospital Triemli, Zurich
  - Klinik Hirslanden, Zurich
  - UniversitaetsSpital Zuerich, Zurich

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Taverna CJ, Baasi S, Hitz F, et al.: First results of long-term rituximab maintenance treatment in follicular lymphoma: safety analysis of the randomized phase III trial SAKK 35/03. [Abstract] J Clin Oncol 27 (Suppl 15): A-8534, 2009.
- [Result] First results of long term rituximab maintenance treatment in follicular lymphoma: safety analysis of the randomized phase III trial SAKK 35/03. F. Hitz, S. Bassi, C. Taverna, W. Mingrone, T. Pabst, L. Cevreska, A. Del Giglio, D.A. Vorobiof, M. Simcock, M. Ghielmini Haematologica (2009) 94: s2; abstract 0413
- [Result] First results of long term rituximab maintenance treatment in follicular lymphoma: safety analysis of the randomized phase III trial SAKK 35/03. C.J. Taverna, S. Bassi, F. Hitz, W. Mingrone, T. Pabst, L. Cevreska, A. del Giglio, D.A. Vorobiof, M. Simcock, M. Ghielmini J Clin Oncol (2009) 27: 15s supplement; abstract 8534
- [Result] Rituximab maintenance treatment for a maximum of 5 years in follicular lymphoma: safety analysis of the randomized phase III trial SAKK 35/03. C. J. Taverna, S. Bassi, F. Hitz, W. Mingrone, T. Pabst, L. Cevreska, A. del Giglio, D.A. Vorobiof, M. Simcock, M. Ghielmini Blood (2010) 116: ASH Annual Meeting abstracts; abstract 1802
- [Result] Taverna C, Martinelli G, Hitz F, Mingrone W, Pabst T, Cevreska L, Del Giglio A, Vanazzi A, Laszlo D, Raats J, Rauch D, Vorobiof DA, Lohri A, Biaggi Rudolf C, Rondeau S, Rusterholz C, Heijnen IA, Zucca E, Ghielmini M. Rituximab Maintenance for a Maximum of 5 Years After Single-Agent Rituximab Induction in Follicular Lymphoma: Results of the Randomized Controlled Phase III Trial SAKK 35/03. J Clin Oncol. 2016 Feb 10;34(5):495-500. doi: 10.1200/JCO.2015.61.3968. Epub 2015 Dec 28. PMID 26712227